CLINICAL TRIAL: NCT01038102
Title: Role of Dietary Fatty Acids in Fatty Liver and Insulin Resistance: a Randomized Controlled Study
Brief Title: Role of Dietary Fatty Acids in Fatty Liver and Insulin Resistance
Acronym: HEPFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Ulf Risérus, Ass. professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAS-2008-1364; CKFUU-45521 (Other Grant/Funding Number: Center for clinical research Dalarna 2009)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2009-12

CONDITIONS: Obesity; Diabetes; Insulin Resistance; Fatty Liver
Keywords: Obesity; Diabetes; Insulin resistance; Fatty liver; NAFLD; Steatosis; Dietary fatty acids
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Insulin Resistance; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PUFA diet (Active Comparator): Diet high in polyunsaturated (rich in linoleic acid, omega-6) fat (15 E%)
  Interventions: Other: PUFA Diet
- SFA diet (Active Comparator): Diet high in saturated fat (15 E%)
  Interventions: Other: SFA diet

INTERVENTIONS:
Other: PUFA Diet — Diet high in polyunsaturated (rich in linoleic acid, omega-6) fat (15 E%).
  Arms: PUFA diet
Other: SFA diet — Diet high in saturated fat (15E%)
  Arms: SFA diet

SUMMARY:
The purpose of this study is to investigate whether substituting saturated fats with polyunsaturated fats reduces fatty liver and improves insulin action and other metabolic variables in abdominally obese subjects

DETAILED DESCRIPTION:
Specific goals:

1. Investigate if substituting saturated fats with polyunsaturated fats reduces steatosis and improves hepatic and/or peripheral insulin action in abdominally obese subjects with type 2 diabetes
2. Investigate if changes of lipogenic enzymes in response to dietary fat intervention are associated with changes in hepatic/peripheral insulin sensitivity or liver fat content
3. Investigate potential mechanism of the effects of dietary fatty acids; e.g. gene expression and lipogenic enzyme activity

ELIGIBILITY:
Inclusion Criteria:

* abdominal obese subjects with or without type 2 diabetes
* sagittal abdominal diameter >25cm

Exclusion Criteria:

* insulin treatment
* history of serious cardiovascular events
* morbid obesity
* claustrophobia (relative criterion)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Hepatic steatosis by MRT | 10 weeks

SECONDARY OUTCOMES:
Insulin resistance by oral glucose tolerance test | 10 weeks
Changes in adipose tissue gene expression and lipogenic enzyme activity | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Risérus, PhD, Principal Investigator — Clinical Nutrition and Metabolism, Dept. of Public Health and Caring Sciences, Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala Science Park, Uppsala, Sweden

REFERENCES:
- [Background] Summers LK, Fielding BA, Bradshaw HA, Ilic V, Beysen C, Clark ML, Moore NR, Frayn KN. Substituting dietary saturated fat with polyunsaturated fat changes abdominal fat distribution and improves insulin sensitivity. Diabetologia. 2002 Mar;45(3):369-77. doi: 10.1007/s00125-001-0768-3. PMID 11914742
- [Background] Yki-Jarvinen H. Fat in the liver and insulin resistance. Ann Med. 2005;37(5):347-56. doi: 10.1080/07853890510037383. PMID 16179270
- [Derived] Bjermo H, Iggman D, Kullberg J, Dahlman I, Johansson L, Persson L, Berglund J, Pulkki K, Basu S, Uusitupa M, Rudling M, Arner P, Cederholm T, Ahlstrom H, Riserus U. Effects of n-6 PUFAs compared with SFAs on liver fat, lipoproteins, and inflammation in abdominal obesity: a randomized controlled trial. Am J Clin Nutr. 2012 May;95(5):1003-12. doi: 10.3945/ajcn.111.030114. Epub 2012 Apr 4. PMID 22492369